CLINICAL TRIAL: NCT06691100
Title: The Acute Effects of an Endurance Exercise Bout the Gut Microbiome and Gut-derived Metabolome in Women's Distinct Fitness and Body Mass Indexes
Brief Title: How a Single Workout Affects Gut Bugs in Women With Different Fitness Levels and Body Types
Acronym: FITGut-W
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCR245983
Record Dates: First submitted 2024-11-12; First posted 2024-11-15 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Weight Management; Obesity; Exercise; Women; Gut Microbiome; Metabolome; Health; Gut Microbiota
Keywords: Gut Microbiota; Womens Health; Exercise; Weight Management; Obesity
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): 30-minute exercise bout in a cycle ergometer at 60 to 70% of the Heart Rate Reserve (HRR) and corresponding power (watts).
  Interventions: Behavioral: Aerobic Exercise

INTERVENTIONS:
Behavioral: Aerobic Exercise — 30-minute exercise bout in a cycle ergometer at 60 to 70% of the Heart Rate Reserve (HRR) and corresponding power (watts).

SUMMARY:
This study aims to elucidate the differences in the gut microbiome functional activity and metabolome in adult premenopausal women with distinctive fitness levels and BMIs (with obesity, w/o obesity). The specific aims are as follows:

* Aim 1: To examine the effects of acute aerobic exercise at 60-70% heart rate reserve (HRRmax) for 30 minutes bout on changes in the abundance of SCFA-producing bacteria and their functional downstream metabolic activity.
* Aim 2: To examine the effects of acute aerobic exercise at 60-70% HRRmax 30-minute bout on changes in GM-released SCFA concentrations in stool and plasmatic metabolome.

DETAILED DESCRIPTION:
Participants who are eligible after completing the online questionnaire will be invited to three in-person visits:

VISIT A (baseline visit)

* Participants will receive oral and written information about the study and be allowed to ask questions.
* Participants will sign the informed consent document.
* Inclusion and exclusion criteria will be reviewed.
* Demographic, health, and lifestyle data will be collected.
* Collection of height and weight.
* Body composition analysis via DXA scan
* Strength test: isometric mid-thigh pull and hand-grip strength test.
* Endurance test: A cardiovascular fitness test using a cycle ergometer will be performed.
* Participants will be provided with a hip accelerometer and at-home stool sample collection kit, and an account will be set up using Cronometer software to track their dietary intake during the study.

At VISIT B (exercise test day), after 7 to 12 days after VISIT A, the following procedures will happen:

* Participants will return a stool sample collected within the past 5 days.
* 7 mL of blood draw
* Performed a 30-minute biking exercise bout at their individually calculated 60 to 70% of the HRR.
* 7 mL of blood draw 3 minutes after the exercise

At VISIT C (24 hours post-exercise), after 24 hours from VISIT B, the following procedures will happen:

* 7 mL blood draw
* Participants will return the accelerometer and the second stool sample collected within the past 24 hours.
* Participants will receive a final report explaining their fitness and body composition results.

Potential Risks There are minimal risks associated with this protocol. This study involves a fitness test, two strength tests, and an acute 30-minute exercise bout. The primary risks associated with this protocol are those related to sample collection, including blood and other biological specimen collection procedures, which are typical procedures in the METLAB. Potential discomforts associated with a blood draw are bruising and possible infections. Risks associated with collecting stool samples are no more than those experienced during regular bowel movements. All participants will undergo a cardiovascular fitness test with potential risks like dizziness, dehydration, muscle soreness, or cardiovascular events. Additionally, those participants in the exercise group will be at risk for minimal risk derived from the exercise training, like muscle sprain. The risk of data confidentiality and security loss will be minimized by reducing exposure to risks. These risks will be presented to volunteers before enrollment during the consent process. For volunteers interested in participating in the study, written, signed consent will be obtained.

Steps taken to minimize risks and to protect subjects' welfare To minimize risks and protect the subjects' welfare, IRB approval and written consent from participants for voluntary participation will be obtained. All participants will be provided with a de-identified study ID for confidentiality. All safety and risk assessments are in place at the laboratory to ensure the participants' risks for participating in an exercise trial. Ongoing monitoring and reporting of any adverse effects will be maintained

Blood collection: The blood collection will take place at the GW Metabolic and Exercise Testing Laboratory (METLAB) and will be performed using aseptic techniques by a trained phlebotomist to minimize any ill effects from all blood draws. Participants will be monitored for potential side effects of blood draws, including dizziness, lightheadedness, and nausea.

Stool Collection: Participants will be provided with a discrete at-home stool collection kit to minimize the potential discomfort that might be caused by the collection of stool samples. Briefly, a pair of gloves, a collection container, packaging, and storage material (e.g., 24-hour ice pack) will be provided.

Cardiovascular fitness test (VO2peak): Performing a cardiovascular fitness test typically involves physical exertion. This is a test performed on a regular basis at METLAB. A trained and qualified research staff member will guide the test and instruct the participant along the way. All minimal risks will be reduced by performing the VO2peak test according to the targeted population (adults with obesity); vital signs, including heart rate and blood pressure, will be monitored, and clear instructions will be provided to ensure proper hydration before the test. Participants will be instructed to warm up and cool down, followed by a post-test evaluation to evaluate any symptoms experienced.

Exercise Training Prescription and Supervised Exercise Bout: Risks of the exercise bout will be minimized by ensuring that all participants meet specific inclusion/exclusion criteria. If fatigue or shortness of breath occurs during exercise sessions, rest will be recommended to allow completion of the prescribed exercise. For muscle soreness, light stretching and hot/cold therapy will be recommended to reduce discomfort, and if needed, over-the-counter pain relievers (e.g., aspirin, acetaminophen, ibuprofen) will be advised unless contraindicated. Some soreness is anticipated during the first few days of the intervention, but due to the low-impact, moderately intense nature of the exercises (e.g., cycling), symptoms are expected to be minor and transient. Although minor to moderate orthopedic injuries may occur, severe injuries are not anticipated given the intensity of the prescribed exercise. A trained research assistant will oversee the exercise bout to ensure the correct intensity and monitor for adverse events. During testing, a CPR/AED-certified research team member will always be present, ensuring participants are not left unaccompanied during exercise testing and cool-down. The GW METLAB is equipped with an AED, and prior to each exercise session, participants will be asked about any health changes that may affect their ability to continue in the study.

Data Confidentiality: Confidentiality of all records is strictly maintained by established procedures. All participants found eligible will be randomly assigned a three-digit participant identification number. All data collected, including blood samples, will be labeled with participant ID numbers and never identifying information. All identifiable participant information, including signed consent forms, will be kept locked in a cabinet and secured in the private office of Dr. Ortega-Santos. PI will store the master key file at GW encrypted servers, to which she will have access. Study personnel will have access only under the supervision and prior approval of PI. All de-identified study data will be collected and managed using REDCap (Research Electronic Data Capture). REDCap is a secure web application designed to support data capture for research studies, providing user-friendly web-based case report forms, real-time data entry validation (e.g., for data types and range checks), audit trails, and a de-identified data export mechanism to common statistical packages (SPSS, SAS, Stata, R/S-Plus). The system was developed by a multi-institutional consortium, which includes GWU, and was initiated at Vanderbilt University. All the de-identified data from sequences.

Reporting of Adverse Events. The PI and study staff are familiar with the policies and procedures of the GWU IRB. During data collection, any reports by participants of minor discomfort or any observations of a potential adverse event, whether obviously directly related to the protocol or not, will be noted and reported to the IRB for a determination regarding whether to submit a formal report. A more serious adverse event will be reported immediately, and precautionary measures will be implemented at that time. The PI will then be responsible for reporting any adverse events to the IRB. The PI and the research assistant will then work to ensure other monitoring and reporting requirements are met as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Biological sex: female
* BMI 19 to 24.99 kg/m2 or BMI 30-40 kg/m2
* Exercisers: Exercise at least 4 times per week for 60 minutes (a total of 240 minutes per week) on a programmed exercise training either on endurance sports (e.g., running, cycling, triathlon), strength (e.g., powerlifting), or team sports (e.g., rugby, football, soccer)
* Non-Exercisers: Sedentary individuals who have not reached the PA guidelines (150 minutes of moderate-intensity physical activity a week, 75 minutes of vigorous-intensity physical activity, or an equivalent combination of moderate and vigorous-intensity physical activity).

Exclusion Criteria:

* Biological sex: male
* BMI < 19 kg/m2 or > 40 kg/m2
* Currently pregnant, < 2 years postpartum, lactating
* Currently taking any herbal, fiber, or prebiotic supplement
* Current or 1-month before the study, taking oral or vaginal antibiotics
* Diagnosed with any gastrointestinal, endocrine, digestive, cancer, or cardiovascular disease.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Sex assigned at birth: Female
Enrollment: 40 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-10-16 (Estimated)

PRIMARY OUTCOMES:
Gut Microbiome Composition | Before the exercise intervention and immediately after the intervention
  Shotgun metagenomics will be used to examine the abundance of specific SCFA-producing bacteria in the stool (e.g., Ruminococcus)
Gut Microbiome Function | Before the exercise intervention and immediately after the intervention
  Shotgun metagenomics will be used to examine the BGCs (i.e., the genes within the microbial genome that dictate gut microbial functionality) to investigate functional downstream metabolic activity.
Plasma Metabolome | Before the exercise intervention, immediately after the exercise intervention, and 24 hours before the intervention
  Gas chromatography and mass spectrometry will be used to measure concentrations of SCFAs in plasma before and after the exercise intervention
Stool Metabolome | Before the exercise intervention, immediately after the exercise intervention, and 24 hours before the intervention
  Gas chromatography and mass spectrometry will be used to measure concentrations of SCFAs in stool before and after the exercise intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Milken Institute School of Public Health, The George Washington University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
We will not be sharing individual participant data (IPD) for this study. Protecting participant privacy is a priority; even de-identified data carries a risk of re-identification, particularly in a smaller sample.

REFERENCES:
- See also: Pre-Screening Survey — https://forms.gle/FdzZdFWSeqT74X949